CLINICAL TRIAL: NCT04426474
Title: A Multiple-Dose Study in Participants With Type 2 Diabetes Mellitus to Investigate the Safety, Tolerability, Pharmacokinetics,and Pharmacodynamics of LY3502970
Brief Title: A Study of LY3502970 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17681; J2A-MC-GZGC (Other: Eli Lilly and Company); 2020-000125-86 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3502970 (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3502970 — Administered orally.
  Arms: LY3502970
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety of LY3502970 and any side effects that might be associated with it. Blood tests will be done to measure how much LY3502970 is in the bloodstream, how long it takes the body to eliminate it, and how it affects blood sugar. Participation could last up to 18 weeks and may include up to 14 visits (including three overnight stays) in the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) for at least 6 months
* Have a glycated hemoglobin (HbA1c) value at screening of greater than or equal to (≥)7.0 percent (%) and less than or equal to (≤)10.5% and are treated with diet and exercise alone or a stable dose of metformin for at least 3 months prior to screening
* Have a body weight of ≥45 kilograms (kg) and have a body mass index of 18.5 to 45 kilograms per square meter (kg/m²), inclusive
* Have had a stable body weight for the 3 months prior to screening (less than [<]5% body weight change)
* Males and females (not considered woman of childbearing potential)

Exclusion Criteria:

* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults or have had an episode of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening
* Have had any of the following within the past 6 months prior to screening: myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischemic attack, cerebrovascular accident or decompensated congestive heart failure, or currently have New York Health Association Class III or IV heart failure
* Show evidence of hepatitis B, and/or positive hepatitis B surface antigen
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Any glucose-lowering medications other than metformin within 3 months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline through Follow-up (up to Day 105)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3502970 | Day 1 through Day 84: Predose up to 96 hours postdose
  PK: Cmax of LY3502970
PK: Area Under the Concentration Versus Time Curve of LY3502970 | Day 1 through Day 84: Predose up to 96 hours postdose
  PK: AUC of LY3502970
Pharmacodynamics (PD): Change from Baseline to Week 12 in Fasting Plasma Glucose (FPG) | Baseline, Week 12
  Pharmacodynamics (PD): Change from Baseline to Week 12 in FPG
PD: Change from Baseline to Week 12 in Fasting Insulin | Baseline, Week 12
  PD: Change from Baseline to Week 12 in Fasting Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (4):
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Hassman Research Institute, Marlton, New Jersey
  - Midwest Clinical Research Unit, Dayton, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas
- Germany (2):
  - Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia
  - Profil Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3502970 in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/7zwMq2LwDbIpQoxy04CHQ7